CLINICAL TRIAL: NCT05332210
Title: A Long-term Open-label Extension Study to Evaluate the Safety of HBM9161 (HL161) Subcutaneous Injection in Patients With Generalized Myasthenia Gravis
Brief Title: Evaluate the Safety of HBM9161 (HL161) Subcutaneous Injection in Patients With Generalized Myasthenia Gravis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9161.7
Record Dates: First submitted 2022-04-06; First posted 2022-04-18 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — HBM9161

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBM9161 Drug Product (680mg) (Experimental): HBM9161 680mg: subcutaneous injection, 6 times per treatment cycle, once a week; the second cycle of treatment may start 4 weeks after the last dose of the previous treatment cycle; if the disease state is still stable 4 weeks after the last dose, the observation can be continued until the disease activity is aggravated (improvement of MG-ADL < 3 points compared with the previous treatment cycle), and the next treatment cycle can start.
  The dose may be reduced to 340 per investigator's discretion. Return to the dose of 680 mg is not permitted after a dose reduction is made.
  Interventions: Drug: HBM9161 Injection (680mg)

INTERVENTIONS:
Drug: HBM9161 Injection (680mg) — HBM9161 Injection

SUMMARY:
The primary study objective is to evaluate medium- and long-term safety of HBM9161 in combination with background treatment for gMG patients through the observation on adverse events and laboratory abnormalities during study period.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the HBM9161.3 Phase 3 study
2. Signed written informed consent.
3. Suitable for continued treatment with HBM9161 as judged by the investigator.
4. Female patients of childbearing potential and male patients with female partners of childbearing potential can participate in this study, but reliable contraceptive measures must be taken (such as physical barrier contraception (patients and their partners), contraceptive pills or patches, spermicide and barrier or intrauterine device). Up to 60 days after the last dose.
5. A negative urine pregnancy at baseline must be observed for women of childbearing age.

Exclusion Criteria:

1. Had received any other clinical study drug since the administration of the study drug in the 9161.3 Phase 3 study.
2. Females who are pregnant or lactating or planning to become pregnant during the study period, or females of childbearing potential who are not using an effective method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs during the study | during the study，up to 24 weeks
  Incidence of AEs

SECONDARY OUTCOMES:
Proportion of patients with sustained improvement | during each treatment cycle (5-week treatment period + 4-week observation period, from the first dose of the cycle to Day 64 of the cycle)
  Sustained reduction defined as MG-ADL score improved by ≥ 3 points from baseline for at least 4 consecutive weeks during the 9-week treatment cycle
During the 24-week study, proportion of time that MG-ADL improved from baseline by 3 or more points | during the study，up to 24 weeks
Proportion of time remained in Minimal Symptom Expression | during the study，up to 24 weeks
  from baseline to Week 24, percentage of time MG-ADL score being 0 or 1
Improvement of patients' quality of life | during the study，up to 24 weeks
  Improvement of patients' quality of life
Incidence and duration of serum anti-HBM9161 antibodies and neutralizing antibodies | during the study，up to 24 weeks
  Incidence and duration of serum anti-HBM9161 antibodies and neutralizing antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China